CLINICAL TRIAL: NCT00745368
Title: Comparing Raltegravir Genital Tract Distribution in HIV-infected Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Robert Dicenzo, Adjunct Assistant Professor of Medicine, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 33113
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Results first posted 2012-10-10 (Estimated); Last update posted 2012-10-10 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections
Keywords: HIV; Raltegravir; pharmacokinetics; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir (Experimental): Raltegravir 400 mg tablets twice daily
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — 400 mg tablets twice daily during duration of trial

SUMMARY:
The purpose of this research study is to determine how much raltegravir gets into the male and female genital tract.

DETAILED DESCRIPTION:
Although we have many medications to fight the HIV virus, very little is known about how much of these medications get into the genital tract. Raltegravir is a new HIV medication that blocks HIV growth and lowers the amount of virus in the blood in a way that is different than all other currently available HIV medications. Raltegravir was recently approved by the Food and Drug Administration (FDA) for use in HIV infected patients, but there is very little information concerning how much raltegravir will reach the genital tract of men or women. The purpose of this research study is to determine how much raltegravir gets into the male and female genital tract.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of blood seropositive for HIV based on self report and confirmed by ELISA and Western blot or detectable HIV RNA

  * Stable anti-retroviral regimen for at least 3 weeks prior to enrollment
  * Capable of giving informed consent
  * Age 18 years and older

Exclusion Criteria:

* Neoplasms
* Women who are pregnant or nursing
* History or current evidence of any significant acute or chronic medical illness that in the opinion of the investigator would preclude the subject from safely participating in the study
* Current use of phenobarbital, phenytoin, or rifampin
* Any major surgery within 4 weeks of enrollment
* Blood transfusion within 4 weeks of enrollment
* Inability to tolerate oral medication
* Inability to tolerate venipuncture, venous access, or genital tract sampling
* History of recent (within 6 months) drug or alcohol abuse
* Evidence of organ dysfunction or any clinically significant deviation from normal in the medical history, physical examination, vital signs, and or clinical laboratory determinations that in the opinion of the investigator would preclude the subject from safely participating in the study
* Any other sound medical, psychiatric and or social reason for exclusion as determined by the investigator
* History of allergy to study medication or related compounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Raltegravir
Started | 19 (Of the 28 subjects who enrolled, 19 participated in a study visit)
Completed | 16 (3 male subjects were unable to provide a sample and are not included in the results)
Not Completed | 3
Not completed — Unable to provide sample | 3

BASELINE CHARACTERISTICS:
Arm/Group | Raltegravir
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Raltegravir Male Genital Tract Concentration
Time Frame: 8-10 hours after raltegravir dose
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Raltegravir
Number analyzed (Participants) | 8
ng/mL | 485.1 [428.5 to 753.3]

2. Primary Outcome: Raltegravir Female Genital Tract Concentration
Time Frame: 8-10 hours after raltegravir dose
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Raltegravir
Number analyzed (Participants) | 8
ng/mL | 879.1 [128.4 to 3541.4]

3. Primary Outcome: Male Paired Plasma Concentration
Description: This sample was taken as close to the time of genital tract sample as possible
Time Frame: 8-10 hours after raltegravir dose
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Raltegravir
Number analyzed (Participants) | 8
ng/mL | 172 [104.3 to 231.0]

4. Primary Outcome: Female Paired Plasma Concentration
Description: This sample was taken as close to the time of genital tract sample as possible
Time Frame: 8-10 hours after raltegravir dose
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Raltegravir
Number analyzed (Participants) | 8
ng/mL | 264.6 [129.4 to 1256.7]

5. Primary Outcome: Male Time Since Last Dose
Description: This measure describes the amount of time that expired between when the dose was administered and when the sample was taken
Time Frame: 8-10 hours after raltegravir dose
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Raltegravir
Number analyzed (Participants) | 8
hours | 8.0 [8.0 to 8.1]

6. Primary Outcome: Female Time Since Last Dose
Description: as for outcome 5
Time Frame: 8-10 hours after raltegravir dose
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Raltegravir
Number analyzed (Participants) | 8
hours | 8.5 [8.2 to 8.6]

7. Primary Outcome: Male Genital Tract:Plasma Concentration Ratio
Description: Units of raltegravir concentration for genital tract and plasma sample are ng/mL
Time Frame: 8-10 hours after raltegravir dose
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Raltegravir
Number analyzed (Participants) | 8
ratio | 4.3 [2.7 to 5.9]

8. Primary Outcome: Female Genital Tract:Plasma Concentration Ratio
Description: Units of raltegravir concentration for genital tract and plasma sample are ng/mL
Time Frame: 8-10 hours after raltegravir dose
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Raltegravir
Number analyzed (Participants) | 8
ratio | 2.2 [0.6 to 5.6]

ADVERSE EVENTS:
Arm/Group | Raltegravir
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
Due to limited sample size and large intersubject variability, more study comparing male and female GT concentrations is needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less